CLINICAL TRIAL: NCT06171126
Title: The Role of Donor Selection on the Outcome of Faecal Microbiota Transplantation (FMT) in Patients With Irritable Bowel Syndrome: a Multi-center Randomised, Double-blinded Placebo-controlled Study
Brief Title: Donor Selection for Faecal Microbiota Transplantation in Irritable Bowel Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 630339
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Fecal microbiota transplantation; Intestinal microbiota; Donor; Dysbiosis; Abdominal symptom; Fatigue; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Dysbiosis; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Own faeces instilled to the small intestine during gastroscopy
  Interventions: Dietary Supplement: Placebo
- Arm A (Experimental): 90g of faeces from Donor A is instilled to the small intestine during gastroscopy
  Interventions: Dietary Supplement: Faeces from donor A
- Arm B (Experimental): 90g of faeces from Donor B is instilled to the small intestine during gastroscopy
  Interventions: Dietary Supplement: Faeces from donor B
- Arm C (Experimental): 90g of faeces from Donor C is instilled to the small intestine during gastroscopy
  Interventions: Dietary Supplement: Faeces from donor C

INTERVENTIONS:
Dietary Supplement: Placebo — By gastroscopy
  Arms: Placebo
Dietary Supplement: Faeces from donor A — By gastroscopy
  Arms: Arm A
Dietary Supplement: Faeces from donor B — By gastroscopy
  Arms: Arm B
Dietary Supplement: Faeces from donor C — By gastroscopy
  Arms: Arm C

SUMMARY:
Five hundred patients are randomized 1:1:1:1 into placebo (own feces), or receiving 90 g fecal transplant from donor A, donor B or donor C. The fecal transplant is administered to the distal duodenum via the working channel of a gastroscope. The patients shall complete 6 questionnaires measuring symptoms, fatigue, quality of life, stool form and diet intake at the baseline and at the end point of the trial and provide a feces sample at the baseline, and at 3, 6 and 12 months after FMT. Dysbiosis and fecal bacterial profile are determined by using 16S rRNA gene PCR DNA amplification/probe hybridization covering regions V3-V9.

DETAILED DESCRIPTION:
Study Description Brief Summary: Five hundred patients are randomized1:1:1:1 into placebo (own feces), receiving 90 g fecal transplant from donor A, donor B or donor C. The fecal transplant is administered to distal duodenum via working channel of a gastroscope. The patients shall complete 5 questionnaires measuring symptoms, fatigue, quality of life and diet intake at the baseline and at the end point of the trial and provide a feces sample at the baseline, and at 3, 6 and 12 months after FMT. Dysbiosis and fecal bacterial are determined by using 16S rRNA gene PCR DNA amplification/probe hybridization covering regions V3-V9.

Detailed Description: Patients: Five hundred patients who fulfil Rome IV criteria for irritable bowel syndrome (IBS) shall be included in the study. All IBS subtypes shall be included with the exception of IBS-U. Donors: The investigators have selected 3 donors (A, B and C) according to the criteria used in their previous randomised double-blind, placebo-controlled study. These criteria included: being a healthy man or woman with no history of disease and no use of medications, aged 20-50 years, being a non-smoker, and exercising regularly. They were borne by vaginal delivery and breastfed. They were treated only a few times with antibiotics during their life. They are screened according to the European guidelines for donors for FMT. Before they are accepted as donors, the bacterial profile and dysbiosis were analysed in a faecal sample using the GA-map dysbiosis test, with a dysbiosis index (DI)= 1, indicating normobiosis. Their feces shall be tested every third month during the trial to exclude communicable disease. Donor A is a male aged 41 years, donor B is a female aged 31 and donor C is a male aged 35.

Protocol: The patients are randomized 1:1:1:1 into placebo (to receive their own feces), to receive 90 g fecal transplant from donor A, from donor B or donor C. Fecal transplant is administered to the distal duodenum via the working channel of a gastroscope. The patients shall complete 5 questionnaires and deliver fecal samples at the baseline, and at 3 , 6 , and 12 months after FMT. Feces collection, preparation and administration: Faeces from both the donors and patients shall be collected and stored at - 80ºC. Frozen donor faeces shall be thawed in the refrigerator at 4ºC, and dissolved in 200 mL of 4ºC cold 0.9% sterile saline. The dissolved stool is administrated to the patients, after an overnight fast, through the working channel of a gastroduodenoscope in the pars descendens of the duodenum always distal to the papilla of Vater. Questionnaires

1. IBS Symptom Severity Scale (IBS-SSS).
2. Birmingham Symptom Scale.
3. Fatigue Assessment Scale (FAS).
4. IBS-quality of life (IBSQoL) Questionnaire.
5. A 5-points subjective global assessment scale
6. Bristol Stool Form Scale

Bacterial analysis: Fecal bacterial analysis is performed using a 16S rRNA gene PCR DNA amplification/probe hybridization technique covering regions V3-V9. DNA extraction is done by using magnetic beads. DI is based on 174 DNA probes targeting more than 300 bacterial strains based on their 16S rRNA sequence in seven variable regions (V3-V9). Probe labelling is by single nucleotide extension and hybridization to complementary probes coupled to magnetic beads, and signal detection by using BioCode 1000A 128-Plex Analyser (Applied BioCode, Santa Fe Springs, CA, USA). A DI above 2 shows a microbiota profile that differs from that of the normobiotic reference collection (DI 1-2: non-dysbiosis, DI: moderate, DI 4-5: severe dysbiosis).

ELIGIBILITY:
Inclusion Criteria:

* Patients who fulfil Rome IV criteria for the

diagnosis of IBS.

* Patients were investigated to exclude other

gastrointestinal organic cause(s).

* Moderate-to-severe IBS symptoms, as indicated

by a score of ≥175 on the IBS-SSS questionnaire

Exclusion Criteria:

* Pregnant, women planning pregnancy or lactating women.
* The use of antibiotics or probiotics within 1

month prior to FMT.

* Having undergone any abdominal surgery, with

the exception of appendectomy, cholecystectomy,

caesarean section and hysterectomy.

* Previous treatment with FMT.
* Immunocompromised patients including those being

treated by immunosuppressive medications.

* Patients with co-morbidity such as kidney failure,

diabetes or chronic heart disease.

* Patients with serious psychiatric disorders

or alcohol or drug abuse.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in IBS-Severity Scoring System total score | 12 months after FMT
  Irritable Bowel Syndrome-Severity Scoring System (IBS-SSS) is a visual analogue scale questionnaire with a total score between 0 and 500 points, with "0" meaning no symptom and higher scores meaning increasing severity. A decrease in total score by ≥50 points is considered as a meaningful response.

SECONDARY OUTCOMES:
Change in dysbiosis index | 12 months after FMT
  Dysbiosis index (DI) is a 5-scale index. A DI above 2 shows a microbiota profile that differs from that of the normobiotic reference collection (DI 1-2: non-dysbiosis, DI 3: moderate, DI 4-5: severe dysbiosis

CONTACTS AND LOCATIONS:
Overall Officials: Jan G Hatlebakk, PhD, Study Chair — Haukeland University Hospital
Locations (3):
- Norway (3):
  - Haukeland University Hospital, Bergen, Vestland
  - Helse Møre og Romsdal HF, Ålesund
  - Diakonhjemmet, Oslo

IPD SHARING:
Plan to Share IPD: Yes
After the completion of the study, study data may be made available to other researchers after contacting the primary investigator
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After completion of the study